CLINICAL TRIAL: NCT05034861
Title: COmputerized CTG Self-MOnitoring Versus Standard Doppler Assessment in Late-onset FGR: Study Protocol for a Randomized Controlled Trial
Brief Title: COmputerized CTG Self-MOnitoring Versus Standard Doppler Assessment in Late-onset FGR: COSMOS Study
Acronym: COSMOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Mother and Child, Warsaw, Poland (Other)
Collaborators: Bielanski Hospital (Other)
Responsible Party: Principal Investigator, Urszula Nowacka, Principal Investigator, Institute of Mother and Child, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: InstituteMCPoland
Record Dates: First submitted 2021-08-13; First posted 2021-09-05 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Fetal Growth Restriction
Keywords: fetal growth restriction; fetal growth retardation; pregnancy; cardiotocography; ultrasound; Doppler; intrauterine growth restriction; maternal-fetal medicine; obstetrics
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Echocardiography, Doppler

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cCTG (Experimental): cCTG group, that will undergo a following process: EFW and Doppler assessment biweekly, and instead of additional weekly Doppler-only assessment, the patients will be provided with an electronic cCTG device at no cost (Carebits). Women will be asked to apply Carebits device at least twice weekly for at least 30 minutes (e.g. Mondays-Thursdays) with minimum 72 hours interval in case of 2 sessions per week. The trace will be examined by an independent centre, available 24 hours daily. The person examining the trace is trained or already specialized in Obs&Gynae. In case of situation requiring medical intervention, the patient will be immediately contacted by phone and advised to self-refer to the nearest Antenatal Unit. In case of normal trace, a full report will follow within 30 minutes after last reading of the trace.
  Interventions: Device: cCTG
- Doppler (Active Comparator): Doppler group, that will undergo a standard process of antenatal care in case of FGR. The EFW and CTG STV will be assessed biweekly. In case of positive end-diastolic flow in UA, Doppler assessment (MCA PI, UA PI, DV PI, Ut PI) will be provided on a weekly basis. In case of deterioration to AEDF/REDF, further management will depend on clinical situation and the patient will be excluded from the study group (applies to both arms).
  Interventions: Diagnostic Test: Doppler

INTERVENTIONS:
Device: cCTG — Self-applied home computerized CTG device used twice weekly instead of standard Doppler assessment once weekly.
  Other Names: Carebits device; www.carebits.pl
  Arms: cCTG
Diagnostic Test: Doppler — Standard Doppler assessment provided once weekly in case of late FGR with positive end diastolic flow in the umbilical artery.
  Other Names: Doppler assessment
  Arms: Doppler

SUMMARY:
Fetal growth restriction is one of the major causes of perinatal morbidity, mortality and adverse neurological outcome. Growth restricted fetuses do not reach their potential due to multiple factors. Although early (<32 weeks' gestation) FGR is associated with the highest risk of adverse outcomes, late FGR (≤ 32 weeks' gestation) is more common in daily maternal-fetal medicine care. Despite its' prevalence, optimal standard for monitoring differs between the centers and may be difficult in case of limited access to advanced perinatal care. We present a protocol for COmputerized CTG Self-MOnitoring versus Standard Doppler assessment in Late-onset FGR (COSMOS) trial, which is a prospective, cross-over, open-label and randomized trial that compares two different protocols for late-onset FGR observation.

All women carrying fetuses with late-onset FGR with positive end-diastolic flow in umbilical artery will be invited to participate in the randomized trial. Patients will be randomly divided into two groups: CTG - a group that will receive electronic device for cCTG home assessment, and Doppler - a group that will be monitored according to standard Doppler velocimetry criteria. Further management will depend on the arm of the study. Pregnancy and neonatal outcomes will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years or older,
* singleton pregnancy,
* ≥32+0 and ≤36+6 weeks' of gestation,
* fluent in Polish or English,
* diagnosed with late-onset FGR based of the Delphi criteria,
* with positive EDF in UA,
* with macroscopically normal fetus on ultrasound assessment.

Exclusion Criteria:

* multiple pregnancy,
* fetal malformations,
* abnormal genetic testing results (if available),
* uncertain pregnancy dating,
* indication for immediate delivery within 48 hours after enrollment,
* preterm prelabour rupture of membranes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant individuals
Enrollment: 150 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Condition at birth | 5 minutes after delivery
  Incidence of Apgar score at 5 min <7 or arterial pH of <7.0 or venous <7.1 or resuscitation (compressions, medications, intubation)
Neonatal Intensive Care Unit admission | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 6 weeks after delivery if discharged earlier
  Incidence any admission to the Neonatal Intensive Care Unit
Brain injury | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 6 weeks after delivery if discharged earlier
  Incidence of Intraventricular haemorrhage (IVH) grade II or above-defined as bleeding into the ventricles; or hypoxic-ischaemic encephalopathy or periventricular leukomalacia or seizures recorded by EEG
Ventilation | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 6 weeks after delivery if discharged earlier
  defined as need of positive pressure (continuous positive airway pressure (CPAP or nasal CPAP) or intubation rate
Respiratory distress syndrome | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 6 weeks after delivery if discharged earlier
  defined as need of surfactant and ventilation as a result of prematurity
Cardiovascular support/treatment | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 6 weeks after delivery if discharged earlier
  Incidence of anaemia-defined as low haemoglobin and/or haematocrit requiring blood transfusion or DIC - disseminated coagulopathy or ductus arteriosus treatment or hypotensive treatment
Neonatal sepsis | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 6 weeks after delivery if discharged earlier
  Incidence of confirmed bacteraemia in cultures or necrotizing enterocolitis
  - Necrotising enterocolitis (NEC)
Retinopathy | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 6 weeks after delivery if discharged earlier
  incidence of retinopathy requiring laser or anti-VEGF administration
Fetal/neonatal death | anytime after the recruitment visit or after delivery before discharge from the hospital or up to 4 weeks after delivery if discharged earlier
  Rate of death in utero or after delivery before discharge from the hospital or up to 4 weeks after delivery if discharged earlier

SECONDARY OUTCOMES:
Maternal anxiety levels | at the recruitment visit and every 2 weeks until delivery
  measured by a screening Generalized Anxiety Disorder 7- question scale (GAD-7 scale). There are four possible answers to all the questions, corresponding to scores 0,1,2,3, respectively, therefore the total score ranges between 0 (not anxious) - 21 (severely anxious).
Compliance | after the recruitment visit until delivery
  adherence to the plan of care - % of the patients attending scheduled visits
Number of hospital visits | after the recruitment visit until delivery
  total number of meetings with the healthcare provider
Mode of delivery | through study completion, an average of 5 weeks after the recruitment visit
  rate of vaginal/caesarean; spontaneous/planned/emergency
Onset of labour | through study completion, an average of 5 weeks after the recruitment visit
  rate of spontaneous/induced/caesarean before uterine contractions
Gestational hypertension | between 20 weeks' gestation - up to 6 weeks after birth
  incidence of new onset hypertension (blood pressure ≥140/90 mmHg) after 20 weeks' of gestation in the absence of preeclampsia as defined by International Society for Study of Hypertension in Pregnancy (ISSHP)
Preeclampsia | between 20 weeks' gestation - up to 6 weeks after birth
  incidence of preeclampsia defined by International Society for Study of Hypertension in Pregnancy (ISSHP) (maternal factors)

CONTACTS AND LOCATIONS:
Overall Officials: Urszula Nowacka, MD, Principal Investigator — Institute of Mother and Child, Warsaw, Poland
Locations (1):
- Institute of Mother and Child, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The deidentified participant data will become available upon publishing the protocol and results of the study. Study protocol will be available immediately following publication.
Access Criteria: The data will be provided on request for anyone after methodologically sound proposal (contact details: urszula.nowacka@imid.med.pl).

REFERENCES:
- [Result] Lees CC, Stampalija T, Baschat A, da Silva Costa F, Ferrazzi E, Figueras F, Hecher K, Kingdom J, Poon LC, Salomon LJ, Unterscheider J. ISUOG Practice Guidelines: diagnosis and management of small-for-gestational-age fetus and fetal growth restriction. Ultrasound Obstet Gynecol. 2020 Aug;56(2):298-312. doi: 10.1002/uog.22134. No abstract available. PMID 32738107
- [Result] Nohuz E, Riviere O, Coste K, Vendittelli F. Prenatal identification of small-for-gestational age and risk of neonatal morbidity and stillbirth. Ultrasound Obstet Gynecol. 2020 May;55(5):621-628. doi: 10.1002/uog.20282. Epub 2020 Apr 6. PMID 30950117
- [Result] Ciobanu A, Khan N, Syngelaki A, Akolekar R, Nicolaides KH. Routine ultrasound at 32 vs 36 weeks' gestation: prediction of small-for-gestational-age neonates. Ultrasound Obstet Gynecol. 2019 Jun;53(6):761-768. doi: 10.1002/uog.20258. Epub 2019 Apr 30. PMID 30883981
- [Result] Figueras F, Gratacos E. Stage-based approach to the management of fetal growth restriction. Prenat Diagn. 2014 Jul;34(7):655-9. doi: 10.1002/pd.4412. Epub 2014 Jun 9. PMID 24839087
- [Result] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Result] Molina LCG, Odibo L, Zientara S, Obican SG, Rodriguez A, Stout M, Odibo AO. Validation of Delphi procedure consensus criteria for defining fetal growth restriction. Ultrasound Obstet Gynecol. 2020 Jul;56(1):61-66. doi: 10.1002/uog.20854. Epub 2020 Jun 7. PMID 31520557
- [Result] Baschat AA. Planning management and delivery of the growth-restricted fetus. Best Pract Res Clin Obstet Gynaecol. 2018 May;49:53-65. doi: 10.1016/j.bpobgyn.2018.02.009. Epub 2018 Mar 1. PMID 29606482
- [Result] Akolekar R, Ciobanu A, Zingler E, Syngelaki A, Nicolaides KH. Routine assessment of cerebroplacental ratio at 35-37 weeks' gestation in the prediction of adverse perinatal outcome. Am J Obstet Gynecol. 2019 Jul;221(1):65.e1-65.e18. doi: 10.1016/j.ajog.2019.03.002. Epub 2019 Mar 13. PMID 30878322
- [Result] Antenatal and postnatal mental health: clinical management and service guidance. London: National Institute for Health and Care Excellence (NICE); 2018 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK553127/ PMID 31990493
- [Result] Lai J, Syngelaki A, Nicolaides KH, von Dadelszen P, Magee LA. Impact of new definitions of preeclampsia at term on identification of adverse maternal and perinatal outcomes. Am J Obstet Gynecol. 2021 May;224(5):518.e1-518.e11. doi: 10.1016/j.ajog.2020.11.004. Epub 2020 Nov 6. PMID 33166504